CLINICAL TRIAL: NCT03145571
Title: Validation of a Midwifery Model in Palestine - Usage and Quality
Brief Title: Validation of a Midwifery Model in Palestine 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Erik Fosse, Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Midwife Palestine
Record Dates: First submitted 2017-04-21; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Maternal Health

STUDY DESIGN:
Intervention Model Description: Specific output monitored in villages where the program had been implemented, and where it was not implemented
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuity of midwifery care (Other): Clinics where the continuity of midwifery care program was implemented during 2013
  Interventions: Procedure: Continuity of midwifery care
- Control (No Intervention): Clinics where no structured changes had been made to the ante- and post- natal care during the period 2013-2015

INTERVENTIONS:
Procedure: Continuity of midwifery care — Pre-natal care in rural villages performed by the midwives from the local hospital
  Arms: Continuity of midwifery care

SUMMARY:
To validate a model of Continuity of Midwifery Care implemented in the region of Nabuls and Jericho in Palestine in 2013, register data from the Palestinian Ministry of Health will be analyzed for the following indicators related to usage and quality.

Changes in these variables before and after the implementation will be compared between the 16 clinics where the model was implemented and all comparable clinics in the region.

DETAILED DESCRIPTION:
In 2013 a program for continuity of midwifery care (midwives at the local hospital provided ante- and post natal care i clinics located in rural villages) in the region Nablus and Jericho on the West Bank, Palestine. By the end of 2013, the model was implemented in 16 of a total of 53 clinics in the region. In order to compare the impact of the continuity of midwifery care on changes in usage of pre- and postnatal services and quality of care, registry data will be obtained from all clinics two years before the implementation (2011-2012) and for two years after the implementation (2014-2015). The following indicators will be compared between the 16 clinics where the program was implemented and comparable clinics where the program has not yet been implemented:

1. Mean number of antenatal visits per woman (Usage primary outcome)
2. Proportion of total pregnant women that visited the clinic (Usage secondary outcome))
3. Percentage of pregnant referred to higher level of care (Quality primary outcome)
4. Percentage of women referred for high blood sugar levels (Quality secondary outcome)
5. Percentage of women receiving postnatal home visits (Quality primary outcome)
6. Proportion of women seen by doctor after birth (Quality secondary outcome)
7. Proportion of newborns seen by doctor after birth (Quality secondary outcome)
8. Total number of consultations for mother and child after birth (Usage secondary outcome)

All data will be obtained from the monthly statistical reports sent from the clinics to the Palestinian Ministry of health.

Data sources, statistical procedures, power and sample size:

The governmental registry includes data from two years before and two years after the implementation. The registry consists of unidentifiable recordings reported monthly from all clinics to the central statistical database in the Ministry of Health. A copy of the heath authority registry was obtained for statistical analysis.

Descriptive and inferential statistics will be used to analyse collected quantitative data. Data will be registered and analysed using the computer statistical package SPSS version 21 and STATA. Prior to analysis all variables will be checked for data file errors.

ELIGIBILITY:
Inclusion Criteria

* All clinics in Nablus and Jericho governorate located in rural areas, that offer pregnancy- and postnatal-care in the whole study period.
* Only clinics that had the intervention continuously during the whole observations period (1st of January 2014 and continued till 31st of December 2015) will be included in the intervention group
* Only the clinics were there were no intervention at all during the whole period will be included in the control group.

Exclusion Criteria:

* Clinics located in urban areas (less than three km from Nablus or Jericho city centre).
* New Clinics that has not been open during the whole study period.
* Clinics were the intervention was only partially implemented

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5760 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Antenatal visits | 0-9 months before delivery
  Mean number of antenatal visits in the clinic per woman

SECONDARY OUTCOMES:
Referral | 0-12 months after delivery
  Percentage of pregnant referred to higher level of care
Home visits | 0-12 months after delivery
  Percentage of women receiving postnatal home visits

OTHER OUTCOMES:
Proportion of visits | 0-9 months before delivery
  Proportion of total pregnant women that visited the clinic
Blood sugar referral | 0-12 months after delivery and 0-9 months before delivery
  Percentage of women referred for high blood sugar levels
Doctor follow-up | 0-12 months after delivery
  Proportion of women seen by doctor after birth
Newborn follow-up | 0-12 months after delivery
  Proportion of newborns seen by doctor after birth
Consultations post partum | 0-12 months after delivery
  Total number of consultations for mother and child after birth

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, MD, PhD, Principal Investigator — Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortensen B, Lukasse M, Diep LM, Lieng M, Abu-Awad A, Suleiman M, Fosse E. Can a midwife-led continuity model improve maternal services in a low-resource setting? A non-randomised cluster intervention study in Palestine. BMJ Open. 2018 Mar 22;8(3):e019568. doi: 10.1136/bmjopen-2017-019568. PMID 29567846